CLINICAL TRIAL: NCT05920993
Title: The Performances and Differences in Tongue Function Between Healthy Adults and Dysphagia in Patients With Stroke in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211024RINC
Record Dates: First submitted 2023-03-06; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-01

CONDITIONS: Cerebrovascular Accident; Healthy Adults
Keywords: tongue strength; healthy adults; tongue function; differences; correlations
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy adults: Measures of tongue function were collected from two groups of individuals(healthy adults and stroke patients with dysphagia ). The items of measurement about healthy adults are the maximal tongue pressure, tongue endurance, and lingual swallowing pressures of saliva, 3-ml water, IDDSI 2, IDDSI3, and IDDSI 4 liquids.
- Stroke patients with dysphagia: The items of measurement about stroke patients with dysphagia are the maximal tongue pressure, tongue endurance, and lingual swallowing pressures of saliva.

SUMMARY:
Cerebrovascular accident makes adults lose the ability to be independent in daily life, and a higher proportion of them will suffer from dysphagia. Previous studies pointed out that the tongue muscle strength of stroke patients is significantly lower than that of healthy adults. Furthermore, the tongue strength of stroke patients with dysphagia is significantly lower than those without dysphagia.

Many studies investigated the performance of tongue function in healthy adults or groups with dysphagia caused by different diseases. However, the current research on the performance of tongue function in healthy adults and stroke patients in Taiwan is relatively lacking. Therefore, our purpose of this study is to investigate the performance and differences of tongue function between healthy adults and strokes patients in Taiwan.

This study is expected to recruit 32 healthy adults and stroke patients in each group. The two groups will be matched with each other by gender and age (±2 years). In the study, Mann assessment of swallowing ability (MASA) will be used as an assessment tool to distinguish whether the subjects are accompany with dysphagia and the severity of dysphagia. And using Iowa Oral Performance Instrument (IOPI) to measure the value of tongue pressure. Then, analyze whether there are significant differences and the correlations. To provide clinicians with empirical data for early detection and intervention of swallowing.

DETAILED DESCRIPTION:
Stroke is one of the causes of disability in adults, and it is easy for patients to lose their ability to be independent in daily life. There are researchers used the Taiwan Stroke Registration Database to investigate the proportion of patients with disability after the first stroke , found that the disability rate was 61.2% one month after stroke, 55.58% after three months, and 51.72% after six months. In addition to changes in consciousness, motor dysfunction, and aphasia, common problems after stroke can also cause dysphagia. Studies have shown that about 51%-55% of patients with acute stroke will be accompanied by dysphagia.

A systematic review showed that patients with dysphagia had a 3-fold higher risk of developing pneumonia (RR=3.17; 95% CI, 2.07, 4.87) than those without 11 times more than those with disabilities (RR=11.56; 95% CI, 3.36, 39.77). Previous study collected the data of 1220 stroke patients in Taiwan from the National Health Insurance Database, divided them into dysphagia group and non-swallowing disorder group, and matched each other by age and sex, and tracked the mortality and aspiration after five years. The incidence of pneumonia, the results of the study showed that after the first year of stroke, the incidence of aspiration pneumonia in the dysphagia group was 4.69 times that of the non-swallowing disorder group, and the five-year mortality rate of the dysphagia group was higher than that of the non-swallowing disorder group 1.84 times. It can be seen that dysphagia has a great impact on stroke patients, even life-threatening.

There are four stages of swallowing, which are the oral preparation stage, oral stage, pharyngeal stage, and esophageal stage. Each stage has its own function, and the tongue plays an important role in the oral stage. It not only provides taste, can also assist chewing, and send the bolus to the pharynx after the bolus is formed, in order to transport the bolus from the oral cavity to the Adequate tongue muscle strength is required in the pharynx, and sufficient tongue muscle strength also prevents vallecular residue after swallowing.

Previous studies have pointed out that the tongue muscle strength of stroke patients is significantly lower than that of healthy adults, and the tongue muscle strength of stroke patients with swallowing disorders is significantly lower than that of stroke patients without swallowing disorders. There are other studies that compare the differences in tongue muscle strength between patients with dysphagia and healthy adults, and even further explore whether there is a cut-off value between the two, so as to provide clinical staff with early detection and intervention for different groups of dysphagia Empirical data.

In order to objectively understand tongue function and strength, many foreign studies have used the Iowa Oral Performance Instrument (IOPI) to explore tongue-related abilities and performance, and to further establish the relationship between tongue muscle strength and tongue endurance in healthy adults. Norm data, and then use this norm to assess whether patients have tongue weakness or as a target reference value for tongue movement planning. In addition to measuring tongue muscle strength and tongue endurance, some scholars also explore the performance of tongue muscle strength when healthy adults swallow liquids of different textures or volumes, as well as dry swallowing and Tongue muscle strength performance when drinking water.

There is a close correlation between muscle strength and skeletal muscle mass, and the reduction of skeletal muscle mass will lead to a decrease in muscle strength, especially after the age of 27, skeletal muscle mass and age begin to show a negative correlation, that is, As a result, skeletal muscle mass gradually decreases with age. In addition to age, skeletal muscle mass also varies with race. Some researchers explored the correlation between race and skeletal muscle mass, pointing out that African Americans have the largest skeletal muscle mass, and then This trend was observed for comparisons of skeletal muscle mass size in Caucasians, Hispanics, and finally Asians, regardless of male or female.

According to past studies on tongue muscle strength, from the same age range and gender, the tongue muscle strength data of healthy adults in different countries are different, which may be caused by racial differences. The data on adult tongue muscle strength and tongue endurance can provide a reference, but considering the differences in race and nationality, it is impossible to apply foreign tongue muscle strength standards to healthy adults in Taiwan. Due to the lack of research data on the tongue function performance of healthy adults and stroke patients in Taiwan, we do not know whether there are differences or correlations between them, nor do we know the physiological values related to different degrees of swallowing disorders and tongue muscle strength What is the relevance of . Therefore, the main motivation of this study is to explore the tongue function performance and differences between healthy adults and stroke patients.

This study aims to investigate the tongue functional performance and differences between healthy adults and stroke patients in Taiwan. On the one hand, we want to understand the functional performance and whether there are differences between the two, as well as the correlation between different degrees of swallowing disorders and tongue pressure measurement items , On the other hand, it also collects tongue performance data in Taiwan to provide clinical personnel as a reference.

The research questions are as follows:

1. In a group of healthy adults, explore the correlation between age and sex and test items.

   (e.g. tongue strength, tongue endurance, the pressure of swallowing saliva, 3-ml water and fluids of varying textures and volumes).
2. In the group of patients with stroke and dysphagia, explore the correlation between age and sex and the test items.

   (e.g. tongue strength, tongue endurance, the pressure of swallowing saliva)
3. To explore the differences between healthy adults and stroke patients with dysphagia in different test items, and whether there is a cut-off value between the two groups (e.g. tongue strength, tongue endurance, the pressure of swallowing saliva)
4. Explore the correlation between the severity of swallowing disorders (mild, moderate, severe) and the test items.

   (e.g. tongue strength, tongue endurance, the pressure of swallowing saliva)

   *The definition of fluids of varying textures: In order to make each texture deployment have a standardized procedure, this research uses International Dysphagia Diet Standardisation Initiative (IDDSI) as the basis for the consistency of the preparation, and the thickener (brand: Neo-High Toromeal) is added to the water as the swallowing food. Using IDDSI level 2 (mildly thick), level 3 (moderately thick), level 4 (pureed) to measure the swallowing tongue muscle strength of healthy adults.

   *The definition of fluids of varying volumes: Divide the volume of each texture into 5ml, 10ml, and 15ml to measure the pressure of tongue muscle of healthy adults in sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dysphagia after stroke:

   * People who recently felt difficulty in swallowing or coughing before/during/after eating or drinking.
   * Over the age of 20
   * Clear consciousness and can complete the following three instructions

     * Is it morning, afternoon or evening?
     * Where is this place?
     * Pease handing me the pen and then point to the ceiling
     * People who have been diagnosed with cerebrovascular disease by a physician
   * MASA total score less than 178 points
2. Healthy adults:

   * People who have not been diagnosed with cerebrovascular disease by a physician
   * Over the age of 20
   * Clear consciousness and can complete the following three instructions

     * Is it morning, afternoon or evening?
     * Where is this place?
     * Pease handing me the pen and then point to the ceiling
     * People who have been diagnosed with cerebrovascular disease by a physician
   * MASA total score is above 178 points

Exclusion Criteria:

* People with a history of neurodegenerative diseases, brain injuries, head and neck cancers, or those who have undergone head and neck surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was divided into two groups, patients with dysphagia after stroke and healthy adults. One group had normal oral motor function, and the other was identified as demonstrating signs of dysphagia caused by cerebrovascular disease. Stroke subjects with dysphagia will be referred by speech-language therapists at National Taiwan University Hospital. Healthy adult subjects will be surveyed by researcher who are age(±2) and sex-matched to stroke patients.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To explore the differences between healthy adults and stroke patients with dysphagia in different test items, and whether there is a cut-off value between the two groups (e.g. tongue strength, tongue endurance, the pressure of swallowing saliva) | up to 3 months
  After completing the above testing items, the statistical method of independent-samples t-test can be used to analyze the data. Based on the analysis results, the numerical values of each observed variable can be compared with the MASA (Modified Ashworth Scale Assessment) scores using Receiver Operating Characteristic (ROC) analysis. Furthermore, the analysis can include the calculation of the Area Under Curve (AUC), sensitivity, specificity, and determination of cut-off points.

SECONDARY OUTCOMES:
In a group of healthy adults, explore the correlation between age and sex and test items. | up to 3 months
  The investigator used the Iowa Oral Performance Instrument (IOPI) to measure the maximum tongue muscle strength in with dysphagia after stroke and healthy adults. The measurement of maximum tongue muscle strength was conducted in peak mode. The examiner placed the tongue pressure bulb on the participant's tongue surface according to the testing sequence and instructed the participant not to move the tongue pressure bulb. Then, the participant was asked to exert maximum upward pressure on the hard palate with their tongue for approximately 2 seconds.
  About the swallowing of saliva and swallowing involves tongue muscle strength with different volumes and textures, the measurement methods and statistical methods used are the same as those for measuring maximum tongue muscle strength.
In the group of patients with dysphagia after stroke, explore the correlation between age and sex and the test items. | up to 3 months
  The investigator used the Iowa Oral Performance Instrument (IOPI) to measure tongue endurance in both with dysphagia after stroke and healthy adults. Tongue endurance was calculated as the duration of time that the participant could sustain 50% of their maximum tongue muscle strength. The duration was measured by the researchers using a stopwatch. The timing started when the pressure reached or exceeded the target pressure (indicated by a green light on the device's panel). However, the timing was stopped if there was a rapid decrease in pressure (when the tongue muscle strength remained between 40% and 50% of the maximum for at least 2 seconds, or if it dropped below 40% for more than 0.5 seconds).
Explore the correlation between the severity of swallowing disorders (mild, moderate, severe) and the test items. | up to 3 months
  To examine the correlation between MASA scores and various observed variables in stroke patients with swallowing disorders, the statistical method of Pearson correlation coefficient can be used. This will help determine the degree of correlation between MASA scores and the different observed variables.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crow HC, Ship JA. Tongue strength and endurance in different aged individuals. J Gerontol A Biol Sci Med Sci. 1996 Sep;51(5):M247-50. doi: 10.1093/gerona/51a.5.m247. PMID 8808997
- [Background] Eltringham SA, Kilner K, Gee M, Sage K, Bray BD, Pownall S, Smith CJ. Impact of Dysphagia Assessment and Management on Risk of Stroke-Associated Pneumonia: A Systematic Review. Cerebrovasc Dis. 2018;46(3-4):99-107. doi: 10.1159/000492730. Epub 2018 Sep 10. PMID 30199856
- [Background] Hirota N, Konaka K, Ono T, Tamine K, Kondo J, Hori K, Yoshimuta Y, Maeda Y, Sakoda S, Naritomi H. Reduced tongue pressure against the hard palate on the paralyzed side during swallowing predicts Dysphagia in patients with acute stroke. Stroke. 2010 Dec;41(12):2982-4. doi: 10.1161/STROKEAHA.110.594960. Epub 2010 Nov 11. PMID 21071718